CLINICAL TRIAL: NCT01034202
Title: A Randomised, Double Blind, Placebo-controlled, Single Dose, Dose-escalating Trial Investigating Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Pegylated Long-acting Human Growth Hormone (NNC126-0083) Compared to Norditropin® SimpleXx® in Healthy Male Subjects
Brief Title: Dose Study in Healthy Males Investigating Safety, Pharmacokinetics and Pharmacodynamics of NNC126-0083 Compared to Norditropin® SimpleXx®
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN8630-1822; 2007-001255-19 (EudraCT Number)
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Growth Hormone Disorder; Healthy
MeSH Terms: interventions — NNC126-0083

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Norditropin® SimpleXx® 0.02 mg/kg + NNC126-0083 (Experimental)
  Interventions: Drug: NNC126-0083; Drug: Norditropin® SimpleXx®
- Norditropin® SimpleXx® 0.04 mg/kg + NNC126-0083 (Experimental)
  Interventions: Drug: NNC126-0083; Drug: Norditropin® SimpleXx®
- Norditropin® SimpleXx® 0.02 mg/kg + placebo (Placebo Comparator)
  Interventions: Drug: placebo; Drug: Norditropin® SimpleXx®
- Norditropin® SimpleXx® 0.04 mg/kg + placebo (Placebo Comparator)
  Interventions: Drug: placebo; Drug: Norditropin® SimpleXx®
- NNC126-0083 (Experimental)
  Interventions: Drug: NNC126-0083
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: NNC126-0083 — One of five dose levels administered subcutaneously (under the skin)
  Arms: Norditropin® SimpleXx® 0.02 mg/kg + NNC126-0083; Norditropin® SimpleXx® 0.04 mg/kg + NNC126-0083
Drug: Norditropin® SimpleXx® — One of two dose levels, followed by NNC126-0083, administered subcutaneously (under the skin)
  Arms: Norditropin® SimpleXx® 0.02 mg/kg + NNC126-0083; Norditropin® SimpleXx® 0.04 mg/kg + NNC126-0083
Drug: placebo — Placebo comparator
  Arms: Norditropin® SimpleXx® 0.02 mg/kg + placebo; Norditropin® SimpleXx® 0.04 mg/kg + placebo; Placebo
Drug: NNC126-0083 — One of three dose levels administered subcutaneously (under the skin)
  Arms: NNC126-0083
Drug: Norditropin® SimpleXx® — One of two dose levels, followed by placebo, administered subcutaneously (under the skin)
  Arms: Norditropin® SimpleXx® 0.02 mg/kg + placebo; Norditropin® SimpleXx® 0.04 mg/kg + placebo

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate the safety, tolerability, pharmacokinetics (exposure of drug) and pharmacodynamics (effect) of NNC126-0083 compared to Norditropin® SimpleXx® and placebo in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smoking male subjects
* Body Mass Index (BMI) between 19.0 and 28.0 kg/m2, both inclusive
* Body weight max. 100 kg

Exclusion Criteria:

* A history or presence of cancer, diabetes, or any clinically significant cardiovascular, respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological, haematological, dermatological, venereal, neurological, psychiatric diseases or other major diseases
* Carrier of Hepatitis B surface antigen (HBsAg) or Hepatitis C antibodies
* Positive result of test for HIV (Human Immunodeficiency Virus) antibodies
* Any clinically significant abnormal haematology or biochemistry screening tests, as judged by the physician
* Clinically significant abnormal ECG (ElectroCardioGram) at screening as evaluated by the physician
* A significant history of alcoholism or drug/chemical abuse, or who has a positive result in the urine drug/alcohol screen, or who consumes more than 28 units of alcohol per week (one unit of alcohol equals about 250 ml of beer or lager, 1 glass of wine, or 20 ml of spirits)
* Habitual smoking, i.e daily smoking or more than 7 cigarettes/week
* Mental incapacity or language barriers which preclude adequate understanding or cooperation, who are unwilling to participate in the trial, or who in the opinion of their general practitioner or the Investigator should not participate in the trial
* Surgery or trauma with significant blood loss within the last 2 months prior to dosing

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2007-08; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | after administration of a single dose of NNC126-0083

SECONDARY OUTCOMES:
Area under the curve (AUC) (0-168h) after a single dose of NNC 126-0083 | 0-168 hours after trial drug administration
Number of injection site reactions | after administration of a single dose of NNC126-0083 and after single dose of Norditropin® SimpleXx®
IGF-I (Insulin-like Growth Factor I) levels | after ascending single doses of NNC126-0083 and a single dose of Norditropin® SimpleXx®

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Hvidovre, Denmark

REFERENCES:
- [Result] Rasmussen MH, Bysted BV, Anderson TW, Klitgaard T, Madsen J. Pegylated long-acting human growth hormone is well-tolerated in healthy subjects and possesses a potential once-weekly pharmacokinetic and pharmacodynamic treatment profile. J Clin Endocrinol Metab. 2010 Jul;95(7):3411-7. doi: 10.1210/jc.2009-2813. Epub 2010 Apr 28. PMID 20427496
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com